CLINICAL TRIAL: NCT03693872
Title: Evaluation of the Nonmotor Symptomatology of Parkinsonian Patients Treated With Two Strategies Related to Apomorphine Pump Therapy in French Hospitals
Acronym: AGAPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 35RC18_9721_AGAPO
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Parkinson Disease
Keywords: Parkinson; Nonmotor symptomatology
MeSH Terms: conditions — Parkinson Disease | interventions — Apomorphine; Dopamine Agonists

STUDY DESIGN:
Intervention Model Description: Interventional to minimal risks and constraints, non randomized, open
Who Masked: Participant
Masking Description: open
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apomorphine (Other): Withdrawal of dopaminergic agonists at pump initiation
  Interventions: Drug: Apomorphine
- Dopaminergic Agonist + Apomorphine (Other): Continuation of dopaminergic agonists at pump initiation
  Interventions: Drug: Dopaminergic Agonist + Apomorphine

INTERVENTIONS:
Drug: Apomorphine — Apomorphine (5 mg/ml), supplied as solution for infusion in a 10 ml glass ampoule Hourly flow rate adjusted during the whole duration of the study to obtain the best effect in each patient
  Other Names: APO
  Arms: Apomorphine
Drug: Dopaminergic Agonist + Apomorphine — Apomorphine (5 mg/ml), supplied as solution for infusion in a 10 ml glass ampoule Hourly flow rate adjusted during the whole duration of the study to obtain the best effect in each patient and associated with dopaminergic agonists
  Other Names: AGAPO
  Arms: Dopaminergic Agonist + Apomorphine

SUMMARY:
There is currently no consensus on the adequate concomitant treatment to apomorphine pump in Parkinson's disease (PD). In practice, some centers withdraw all dopaminergic agonists when initiating apomorphine pump therapy, whereas others combine the two. To date, there has been no study led to determine the best strategy for efficiently treating motor and nonmotor symptoms, as well as improving patients' quality of life (QoL). This preliminary study, entitled AGAPO, aims at identifying significant differences in patients' evolution (nonmotor symptoms and quality of life), over a course of 6 months, depending on the two strategies adopted in French centers (apomorphine pump with or without dopaminergic agonists), through the Non Motor Symptoms Scale (NMSS, Chaudhuri et al, 2017).

DETAILED DESCRIPTION:
The recruitment period will be 24 months. The duration of the study will be 6 months for each patient due to adjustments of apomorphine pump parameters and oral medication as well time needed for motor and nonmotor changes to develop and influence QoL.

This study will be done without any modification of the planned treatment plan for each patient included. The treatments are administered in accordance with their marketing authorization and according to the usual practices of each center. No additional visits are expected.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged = or > 18 years,
* Idiopathic PD (According to British Brain Bank Criteria) without any other known or suspected cause of symptoms,
* Indicated for apomorphine pump therapy and according to the centers' practice, treatment with apomorphine pump association with dopamine agonists or apomorphine pump therapy alone
* Presence of fluctuations for > 3 years,
* Patients covered with social insurance.
* Written informed consent

Exclusion Criteria:

* Neurological (other than Parkinson's disease) or severe psychiatric history (depression, schizophrenia, addiction, bipolar disorder, anxiety and depressive disorders);
* Severe neurocognitive disorders (DSM-V)
* History of use of apomorphine pump treatment or deep brain stimulation or lesional surgery for PD or intrajejunal L-Dopa;
* History or current drug or alcohol abuse or dependencies;
* History of impulse control disorders;
* Adults legally protected (under judicial protection, guardianship or supervision), persons deprived of their liberty;
* Inability to understand the information given on the study, to express informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-06-02 (Actual)

PRIMARY OUTCOMES:
Difference in the Non Motor Symptoms Scale (NMSS) between the Baseline assessment and the assessment at 6 months' follow up | 6 months
  The Non-Motor Symptoms Scale (NMSS) measures the frequency and severity of a range of non-motor symptoms in Parkinson's Disease, through 30 questions grouped into 9 domains: cardiovascular, sleep/fatigue, mood/cognition, perceptual problems/hallucinations, attention/memory, gastro-intestinal tract, urinary, sexual function, and miscellaneous (pain, taste/smell, weight change, excessive sweating). Severity is rated on a scale from 0 (none) to 3 (severe). Frequency is rated on a scale from 1 (rarely) to 4 (very frequent). Item scores are calculated as the product of severity and frequency; the total score is obtained by summing the item scores. The NMSS total score ranges from 0 to 360 with a lower score indicating fewer symptoms. A negative change from baseline indicates improvement in symptoms (reduced score).

SECONDARY OUTCOMES:
Change in the Parkinson's Disease Quality of Life Questionnaire (PDQ39) between the Baseline assessment and the assessment at 6 months' follow up | 6 months
  Parkinson's Disease Quality of Life Questionnaire (PDQ-39): the 39-Item Parkinson's Disease Questionnaire (PDQ-39) is a commonly used measure of self-appraisal in PD. It is a measure of health status and quality of life, by assessing difficulties in 8 dimensions of daily living: mobility (10 items), activities of daily living (6 items), emotional well-being (6 items), stigma (4 items), social support (3 items), cognition (4 items), communication (3 items) and bodily discomfort (3 items). The frequency of each event is determined by selecting one of 5 options: never (scored 0) / occasionally (scored 1) / sometimes (2) / often (3) / always (4). Each dimension total score range from 0 to 100, with lower scores reflecting better quality of life.
Change in the Neurologist Global Impression of change (CGI) between the Baseline assessment and the assessment at 6 months' follow up | 6 months
  The Change in the Neurologist (clinician) Global Impression of change (CGI) provides a brief, stand-alone assessment of the clinician's view of the patient's global functioning prior to and after initiating a study medication. It ranges from severely impaired to dramatically improved.
Change in non-motor aspects of experiences of daily living (MDS-UPDRS I) between the Baseline assessment and the assessment at 6 months' follow up | 6 months
  The Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) is the standard validated tool for the assessment of patients with Parkinson's Disease (PD). This combined scale includes subsections collecting data regarding: nonmotor experiences of daily living (part I), their motor experiences of daily living (part II) an examination of the motor features of PD (part III), and motor complications arising from the use of dopamine replacement (part IV). The Part I include 13 items (6 semistructured interview items and 7 self-reported items) scored on a scale from 0 (normal) to 4 (severe). Higher scores reflect worse condition.
Change in apathy assessed on the long version of Lille Apathy Rating Scale between the Baseline assessment and the assessment at 6 months' follow up (LARS) | 6 months
  The Lille apathy rating scale (LARS) is a measure of apathy through nine domains (each corresponding to a clinical manifestation of apathy: everyday productivity, interests, taking the initiative, novelty seeking, motivation - Voluntary actions, emotional responses, concern, social life & self-awareness) and 33 queries. The interview is structured, with a precise scoring mode for each reply (-2 to 2); when an item does not apply to the patient or the reply cannot be classified, it is scored "0" (for non-applicable and/or non-classifiable) The scale's overall score ranges from -36 to +36, with highest scores reflecting apathy severity. 4 factorial sub-scores (intellectual curiosity, emotion, action initiation and self-awareness) are calculated from sub-scale scores.
Change in occurrence of anxiety (STAI-YA) between the Baseline assessment and the assessment at 6 months' follow up | 6 months
  Present feelings
Change in occurrence of anxiety (STAI-YB) between the Baseline assessment and the assessment at 6 months' follow up | 6 months
  General feelings
Change in behavioral symptoms assessed by Ardouin Scale between the Baseline assessment and the assessment at 6 months' follow up | 6 months
  Changes from baseline in hyper and hypo dopaminergic symptoms scores will be assessed through the Ardouin Scale of Behavior in Parkinson's Disease (ASBPD). It is designed for assessing mood and behavior with a view to quantifying changes related to Parkinson's disease, to dopaminergic medication, and to non-motor fluctuations. Its 21 items address nonmotor symptoms and are grouped into four dimensions: general psychological assessment, apathy, nonmotor fluctuations and hyperdopaminergic behaviors, with a 5-point rating scale ranging from 0 (Absent) to 4 (Severe). A score ≥ 2 is considered as a warning sign.
Change in emotional function assessed by the short form of the TEIQue between the Baseline assessment and the assessment at 6 months' follow upscale | 6 months
  The Trait Emotional Intelligence Questionnaire-Short Form (TEIQue-SF) aims at evaluating emotional intelligence through a self-report inventory that measure global trait emotional intelligence (trait EI) through a 30-item questionnaire. The trait EI is about perceptions and not about abilities, competencies or skills ; high scores are not necessarily adaptive (good) and low scores are not necessarily maladaptive (bad).
Change in emotional function assessed by the short form of the BEQ scale between the Baseline assessment and the assessment at 6 months' follow up | 6 months
  The Berkeley Expressivity Questionnaire (BEQ) is a self-report measure of three emotional expressivity facets related to emotional expressivity: expressivity of negative and positive emotions, and strength of expression impulse. Each of the 16 items is answered on a 7-point Likert-type ranging from 1 (strongly disagree) to 7 (strongly agree). The 3 facets can be kept as separate scores or combined to form an overall Emotional Expressivity score.
Change in motor aspects of experiences of daily in "on" and "off" medication (MDS-UPDRS II) between the Baseline assessment and the assessment at 6 months' follow up | 6 months
  The Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) is the standard validated tool for the assessment of patients with Parkinson's Disease (PD). This combined scale includes subsections collecting data regarding: nonmotor experiences of daily living (part I), their motor experiences of daily living (part II) an examination of the motor features of PD (part III), and motor complications arising from the use of dopamine replacement (part IV). The Part II include 13 self-reported items) scored on a scale from 0 (normal) to 4 (severe). Higher scores reflect worse condition.
Change in motor examination during "on" periods (MDS-UPDRS III) between the Baseline assessment and the assessment at 6 months' follow up | 6 months
  The Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) is the standard validated tool for the assessment of patients with Parkinson's Disease (PD). This combined scale includes subsections collecting data regarding: nonmotor experiences of daily living (part I), their motor experiences of daily living (part II) an examination of the motor features of PD (part III), and motor complications arising from the use of dopamine replacement (part IV). The Part III include 18 items scored on a scale from 0 (normal) to 4 (severe). Higher scores reflect worse condition.
Change in motor complications with MDS-UPDRS IV between the Baseline assessment and the assessment at 6 months' follow up | 6 months
  The Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) is the standard validated tool for the assessment of patients with Parkinson's Disease (PD). This combined scale includes subsections collecting data regarding: nonmotor experiences of daily living (part I), their motor experiences of daily living (part II) an examination of the motor features of PD (part III), and motor complications arising from the use of dopamine replacement (part IV). The Part IV include 6 items assessed in a semistructured interview, scored on a scale from 0 (normal) to 4 (severe). Higher scores reflect worse condition.
Change in motor examination with the Schwab and England scale between the Baseline assessment and the assessment at 6 months' follow up | 6 months
  The Schwab & England activities of daily living evaluates patients' autonomy through a percentage ranging from 0% (=Vegetative functions such as swallowing, bladder and bowel functions are not functioning. Bedridden.) to 100% ( = Completely independent. Able to do all chores without slowness, difficulty or impairment. Essentially normal).
  Unaware of any difficulty.
Change in motor examination with the Hoehn & Yarr scale | 6 months
  The severity of PD is assessed through the Modified Hoehn & Yahr rating scale, consisting of 10levels comprised between 0 (best), 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5 (worst).
Change in cognitive function assessed by the MoCA scale between the Baseline assessment and the assessment at 6 months' follow up | 6 months
  The Montreal Cognitive Assessment (MoCA) is a short tool (one-page 30-point test administered in approximately 10 minutes) to evaluate a multitude of cognitive domains (visuospatial / executive functioning, object naming, memory, attention, language, abstraction, orientation). MoCA scores range between 0 and 30; a score ≥ 26 is considered to be normal.
Change of dose for treatments assessed by levodopa (L-DOPA) équivalents between the Baseline assessment and the assessment at 6 months' follow up | 6 months
Frequency, type and severity of therapy-related adverse events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marc VERIN, PH, Principal Investigator — Rennes University Hospital
Locations (6):
- France (6):
  - Hôpital Gui de Chauliac, Montpellier
  - CH Caremeau, Nîmes
  - CHU La Pitié Salpêtrière, Paris
  - CHU de Reims- hôpital Maison Blanche, Reims
  - CHU de Rennes, Rennes
  - CHU Charles Nicolle, Rouen

IPD SHARING:
Plan to Share IPD: No